CLINICAL TRIAL: NCT06014567
Title: Characterising Biomarkers of Disease and Ageing in Twins Using Magnetic Resonance Imaging
Brief Title: Twins MR Imaging Study
Status: Enrolling by invitation | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 322446
Record Dates: First submitted 2023-07-04; First posted 2023-08-28 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-07

CONDITIONS: Aging
Keywords: Magnetic resonance imaging (MRI); Twins
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — 1. A single (≤45 minutes) brain MRI will include T1w and T2w imaging to assess the morphology and structure of the brain, as well as inflammatory processes. Diffusion-weighted imaging will be used to gain information about internal brain connectivity related to brain functions. MRI, MR angiography (MRA) and fMRI pulse sequences will also be acquired to detect vascular pathologies and brain lesions. T2w morphological images of the whole spine will also be obtained.
  2. A single (≤45 minutes) MR imaging investigation to include cardiovascular, abdominal, and musculoskeletal regions. MRI will be performed to assess the structure and function of these body regions and organs, including functional imaging of the heart. These investigations will include T1w and T2w imaging to assess morphology and structure, mapping studies of T1, T2 and T2*, perfusion imaging and cine imaging to assess the heart dynamically.

SUMMARY:
This study aims to create a comprehensive Magnetic Resonance Imaging data resource in twins aged 18 years and older. The data will be used alone or in conjunction with existing data to explore organ-specific ageing and twin-pair differences related to ageing and disease.

DETAILED DESCRIPTION:
BACKGROUND Diverse interactions between environmental, genetic, and epigenetic factors shape individual paths of ageing and disease. In young adulthood, twins are highly similar in most organ structures, but their similarity decreases over time as they are progressively exposed to different environments. Twin studies provide an ideal way to investigate how the body ages and how age-related diseases (such as Alzheimer's disease, heart failure, fatty liver disease, and cancer) develop. Magnetic Resonance Imaging (MRI) is a type of scan that produces detailed images of the inside of the body. MRI enables non-invasive and safe visualisation of age and disease-related changes in the body, often long before clinical symptoms are perceived. MRI-derived biological features/biomarkers can be used to understand the influence of environmental exposures on ageing and disease.

PARTICIPANTS 2500 adult (age 18 and older) volunteers of TwinsUK, the UK's largest adult twin Biobank and the most clinically detailed globally, will be invited to participate. Interested individuals will complete screening to confirm study eligibility and their safety for MRI scanning. Eligible participants will complete informed consent prior to undertaking research MRI scans of their brain, spine, heart, abdomen and parts of their skeleton and muscles. 350 twins with differences in their data will be invited to repeat the MRI scans about two years later to explore longitudinal multi-organ imaging correlates of key environmental exposures based on cross-sectional signals and existing literature.

PROCEDURES Two 45-minute MRI scans of (1) the head and spine and (2) the abdomen to the upper thigh.

OUTCOMES Imaging-derived measures of morphology and function of the brain, spine, abdominal organs and musculoskeletal tissue. These measures will be used to identify twin pair differences related to ageing and disease. A comprehensive repository of MRI data will be created using protocols harmonised with the UK biobank. This will facilitate subsequent linkage with concurrently acquired samples and historic exposome data in longitudinal twin cohort.

ELIGIBILITY:
Inclusion Criteria:

* Identical or non-identical twins
* Gender: Male or Female
* Age: 18 years or above at the time of recruitment
* Must be able to understand the study information and provide informed consent
* Participation in the TwinsUK Biobank

Exclusion Criteria:

* Pregnancy
* Unable to tolerate MRI Procedures, e.g., claustrophobia, severe anxiety
* Contraindication to MRI Scanning, e.g., presence of non-MR conditional implants
* Any additional condition declared voluntarily by the participant that the principal investigator (PI) deems likely to affect the study's outcome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: TwinsUK Biobank longitudinal registry twin volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
BrainAGE score | At time of scan (duration 45 mins)
  BrainAGE will be calculated using MRI-derived phenotypes of brain volumetric changes (Cole et al, 2017).
BodyAGE score | At time of scan (duration 45 mins)
  BodyAGE will be calculated using MRI-derived phenotypes of organ and tissue changes in the heart, liver, pancreas, kidneys, spine and muscle (Linge et al, 2018).

CONTACTS AND LOCATIONS:
Overall Officials: Claire Steves, Study Chair — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Access to the data may be requested by application to the TwinsUK Resource Executive Committee (TREC).
Supporting Information: Study Protocol, ICF
Time Frame: The data will be available after the primary analyses have been reported and as determined by TREC based on the application data sharing policies. The data will remain available for the foreseeable future with no end date, at present
Access Criteria: See the information in the link.
URL: https://twinsuk.ac.uk/resources-for-researchers/our-data.

REFERENCES:
- [Background] Cole JH, Poudel RPK, Tsagkrasoulis D, Caan MWA, Steves C, Spector TD, Montana G. Predicting brain age with deep learning from raw imaging data results in a reliable and heritable biomarker. Neuroimage. 2017 Dec;163:115-124. doi: 10.1016/j.neuroimage.2017.07.059. Epub 2017 Jul 29. PMID 28765056
- [Background] Linge J, Borga M, West J, Tuthill T, Miller MR, Dumitriu A, Thomas EL, Romu T, Tunon P, Bell JD, Dahlqvist Leinhard O. Body Composition Profiling in the UK Biobank Imaging Study. Obesity (Silver Spring). 2018 Nov;26(11):1785-1795. doi: 10.1002/oby.22210. Epub 2018 May 22. PMID 29785727